CLINICAL TRIAL: NCT07158775
Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of Intravitreal Administration of BS01, a Recombinant Adeno-Associated Virus Vector Expressing ChronosFP (AAV2-CAGChronosFP) in Patients With Geographic Atrophy Secondary to Dry AMD
Brief Title: A Phase 1/2 Study to Evaluate the Safety and Efficacy of Intravitreal Administration of BS01 in Patients With Geographic Atrophy Secondary to Dry AMD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionic Sight LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BS01-GA-001
Record Dates: First submitted 2025-09-04; First posted 2025-09-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy (GA) Secondary to Dry Age-related Macular Degeneration (AMD)
Keywords: GA
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Part 1 is an open label dose-escalation study; Part 2 is a randomized sham-controlled study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BS01 (low dose) (Experimental)
  Interventions: Biological: BS01
- Sham control (Sham Comparator)
  Interventions: Other: Sham procedure control
- BS01 (high dose) (Experimental)
  Interventions: Biological: BS01

INTERVENTIONS:
Biological: BS01 — a recombinant adeno-associated virus vector expressing ChronosFP (AAV2-CAGChronosFP)
  Arms: BS01 (high dose); BS01 (low dose)
Other: Sham procedure control — Sham procedure without needle
  Arms: Sham control

SUMMARY:
This is a Phase 1/2 study, multi-center, dose-escalation interventional study of BS01 in subjects with GA secondary to dry AMD. Part 1 is an open label dose-escalation study; Part 2 is a dose-expansion study with dose(s) selected from Part 1 based on a benefit/risk assessment, and an untreated (sham injection) group to allow for a controlled comparison of efficacy and safety.

This is a seamless Phase 1/2 study in up to 10 patients for Phase 1 and 30 patients Phase 2 in patients with GA secondary to dry AMD.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Signed informed consent obtained before screening.
2. Men or women between 50 and 85 years of age inclusive at the time of signing the informed consent.

Ophthalmic Inclusion Criteria

1. Geographic atrophy with some macula foveal involvement secondary to dry AMD.
2. Total GA area ≥ 5 and ≤ 17.5 mm2 (2 and 7 disk areas respectively), based on Heidelberg Region Finder or equivalent automated software.
3. If GA is multifocal, at least one focal lesion should measure ≥ 1.25 mm2 (0.5 disk area) to ensure measurable focal effects for efficacy evaluation.
4. Composite lesion encompassing confluent GA regions with total area meeting thresholds given in 2 above.
5. GA in part within 1200 microns from the foveal center.
6. The atrophic lesion must be able to be photographed in its entirety.
7. BCVA between 20/50 to 20/400, inclusive, using letter score per EDTRS chart.
8. Clear ocular media and adequate pupillary dilatation in both eyes to allow for all imaging procedures, including good quality stereoscopic fundus photography and fundus autofluorescence (FAF).
9. Central fixation.

Exclusion Criteria:

General Exclusion Criteria

1. Previous therapeutic radiation in the region of the SE.
2. Previous treatment with any ocular or systemic gene transfer product.
3. Any treatment with an investigational agent in the past 60 days for any condition.
4. Women who are pregnant or nursing.
5. Known hypersensitivity to topical ocular anesthetics or diagnostic drops to be used during the study.
6. Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.

Ophthalmic Exclusion Criteria

1. > 30% difference of BCVA using EDTRS in two baseline visual acuity assessments with at least 14 days apart during screening.
2. Any intraocular surgery or thermal laser within 3 months of study entry. Any prior thermal laser in the macular region, regardless of indication.
3. Any ocular or periocular infection (including blepharitis), or ocular surface inflammation in the past 12 weeks.
4. History of any of the following procedures: Posterior vitrectomy, filtering surgery (e.g., trabeculectomy), glaucoma drainage device, corneal transplant, or retinal detachment.
5. Any sign of diabetic retinopathy in either eye.
6. Intraocular pressure (IOP) > 25 mmHg in either eye.
7. Completely atrophic centrally located lesions based on ellipsoid zone (EZ) loss in spectraldomain optical coherence tomography (SD-OCT).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
[Phase 1] Number of the dose limiting toxicities (DLTs), incident and severity of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 12 months
[Phase 2] Change from baseline in BCVA (Best Corrected Visual Acuity) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- NJ Retina, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided